CLINICAL TRIAL: NCT06038175
Title: Is Video Head Impulse Testing a Safe, Reliable and Cost Effective Method of Assessment of Patients Presenting for Dizziness at a Comprehensive Stroke Center?
Brief Title: vHIT Testing for Presentation of Dizziness at a Comprehensive Stroke Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Christine Holmstedt, PI, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Pro00129771
Record Dates: First submitted 2023-09-01; First posted 2023-09-14 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Stroke, Acute; Vertigo; Vertigo, Peripheral; Dizziness; Dizziness; Syndrome
MeSH Terms: conditions — Stroke; Vertigo; Dizziness; Syndrome

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The clinician performing the vHIT will be blinded to the result of the CT scan before entering their report.
  The neurotologist reviewing the results of vHIT testing will be blinded to the patient's presentation, neurologic testing, and CT scan results.
  the clinician performing the vHIT and the neurotologist reviewing the results of vHIT testing are both members of the Study Team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vHIT testing (Experimental): For the research portion of this study, following standard of care examinations listed above, the patient would have a vHIT headset placed on their head for approximately 3-5 minutes to test if they exhibit corrective saccadic movements and to measure gain reduction to identify vestibular hypofunction. During vHIT testing a commercially available mono-ocular video oculography system will be donned on the patient. Subjects will be instructed to maintain fixation at a target from 1 m distance. A study team member will deliver at least 5 head impulses per side in the horizontal and vertical planes with unpredictable timing and direction. A neurotologist will then evaluate the VOR gain or the ratio of eye velocity over-head velocity. The presence of refixation (catch-up) saccades, either overt or covert, will be evaluated by the study team. In line with previous literature, the vHIT testing will be considered to be abnormal if VOR gain is <0.8 in the presence of refixation saccades .
  Interventions: Device: Video Head Impulse Testing; Other: Standard of care neurologic evaluation
- Standard of Care (Active Comparator): The intervention group will be compared to standard of care provided to patients currently admitted for dizziness. Standard of care includes National Institute of Health Stroke Scale evaluation, evaluation by a neurologist, and a CT scan or MRI if warranted.
  Interventions: Other: Standard of care neurologic evaluation

INTERVENTIONS:
Device: Video Head Impulse Testing — During vHIT testing a commercially available mono-ocular video oculography system will be donned on the patient. (Interacoustics EyeSeeCam vHIT 3rd Generation Tests: VOR of lateral, RALP, & LARP canals. SW: 3rd generation VE525 software. HW: laptop PC, lightweight monocular video goggles). Subjects will be instructed to maintain fixation at a target from 1 m distance. A study team member will deliver at least 5 head impulses per side (10-20° angle, duration 150-200 ms, peak velocity of >150°/s) in the horizontal and vertical planes with unpredictable timing and direction. A neurotologist will then evaluate the VOR gain or the ratio of eye velocity over-head velocity. The presence of refixation (catch-up) saccades, either overt or covert, will be evaluated by the study team. In line with previous literature, the vHIT testing will be considered to be abnormal if VOR gain is <0.8 in the presence of refixation saccades .
  Arms: vHIT testing
Other: Standard of care neurologic evaluation — A standard neurologic evaluation will be performed including a National Institute of Health Stroke Scale and imaging if symptoms and NIHSS warrant.

SUMMARY:
The purpose of this study is to evaluate the sensitivity and specificity of the video head impulse test (vHIT) device, when implemented in the acute ED setting to identify acute ischemic stroke or central pathology vs peripheral vestibular dysfunction in patient's presenting with vertigo. This study will evaluate the implementation of the device, consistency with current diagnostic standards, unnecessary administration of antithrombolytics and will further study the reduction in hospital admissions and overall healthcare costs.

DETAILED DESCRIPTION:
In the proposed study, subjects admitted to the Emergency Department (ED) with symptoms of dizziness, concerning for an acute ischemic stroke, will undergo routine triage (bedside neurologic examination, head impulse testing, CT scan) and will then be tested with a vHIT device to attempt to further identify the cause of dizziness, after standard of care testing has been performed. The clinician performing the vHIT will be blinded to the result of the CT scan before entering their report.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18-90
* Admitted to the MUSC ED with symptomatic dizziness, concerning for a stroke vs peripheral vestibular dysfunction.

Exclusion Criteria:

* Prisoners
* COVID +
* Cognitively Impaired Individuals

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity & Specificity of vHIT device | This will be performed once all results are compiled, not to exceed 90 days after study completion.
  Sensitivity and specificity of the vhit to detect peripheral vestibular dysfunction in an acute presentation of vertigo

SECONDARY OUTCOMES:
Time to perform testing | From time the study team member arrives to patient's location until vHIT testing is complete, not to exceed 1 hour.
  The time it takes to perform vHIT testing on a participant admitted for dizziness in the hospital environment.
Predictive Value | At the time results are compared from vHIT testing to CT scan, not to exceed 30 days post testing.
  We will measure positive predicitive value of vHIT to determine peripheral vestibular involvement in a participant who presents with dizziness.
Cost Analysis | This will be performed once all results are compiled, not to exceed 90 days after study completion.
  We will examine the cost reduction that would have occured if vhit was incorporated in decision making for stroke workup and/or hospital admission

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No